CLINICAL TRIAL: NCT06950892
Title: Remote Sputum Collection in Adults With Cystic Fibrosis
Brief Title: Remote Sputum Collection in Cystic Fibrosis
Acronym: RESCUe
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 857045
Record Dates: First submitted 2025-03-27; First posted 2025-04-30 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis; Infections
Keywords: Cystic Fibrosis; Pseudomonas aeruginosa
MeSH Terms: conditions — Cystic Fibrosis; Infections; Pseudomonas Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with cystic fibrosis: People with cystic fibrosis age 18 years or older without a history of solid organ transplantation.

SUMMARY:
Elexacaftor/Tezacaftor/Ivacaftor or Trikafta improves lung health in people with cystic fibrosis (CF), including decreased cough and mucous production. Diagnosing lung infections has become more challenging due to the decrease in sputum and rise of telehealth services. While the option of collecting sputum samples at home and sending them by mail may be feasible, uncertainty remains about how the collection of samples outside of clinic and delays in testing while in the mail impact infection detection. This study will compare bacterial cultures using sputum samples collected at home versus samples collected in clinic (saline-induced sputum and throat swab). This study seeks to shed light on how valuable home collected samples can be and help us better understand the usefulness of home-collected sputum samples for both clinical and research purposes.

DETAILED DESCRIPTION:
The clinical standard of care of people with CF is conducting sputum culture for infection surveillance and detection. However, the introduction of Elexacaftor/Tezacaftor/Ivacaftor (ETI) and adoption of telehealth encounters have reduced the number of respiratory cultures and shifted the types of respiratory sampling over the past three years. People with CF on ETI who were previously able to expectorate sputum are now less likely to produce sputum during clinic visits. As a result, there has been an increase in oropharyngeal (OP) swab sampling in adults. OP swabs lack sensitivity for bacterial detection. Despite clinical improvements related to ETI use (eg lung function, decreased pulmonary exacerbation rates), chronic bacterial infection persists in CF airways. Therefore, additional non-invasive methods for infection surveillance are needed. The investigators propose remote collection of sputum is a promising option for detecting bacteria and fungi in people with CF. Yet, delayed processing and temperature storage conditions may impact the recovery of CF pathogens in remotely collected sputa. To address this, the investigators propose an observational study testing the accuracy and validity of remotely collected sputum. The study will achieve this by comparing CF pathogen detection by culture in sputum samples collected at home to those obtained through induced sputum and OP swabs during clinic visits. The aims of the study are to:

1. Determine the diagnostic performance of home-collected sputum samples for CF pathogen detection compared to clinic-based induced sputum collection.
2. Determine if CF pathogen detection is greater in home-collected sputum compared to OP swab sampling.
3. Determine if storage temperature conditions (ambient versus 4°C) during overnight shipping influence bacterial identification and abundance in home-collected sputum.

The study will enroll 150 participants. The sensitivity, specificity, overall accuracy, positive predictive value (PPV), and negative predictive value (NPV) with 95% confidence intervals will be calculated for the home-collected sputum method and clinic-induced sputum culture performed the local clinical laboratory as the gold standard (Aim 1). A receiver operating characteristic (ROC) curve will be plotted and area under the curve (AUC) will be calculated. Similar analyses will be conducted for Aim 2 using OP swab as the clinical gold standard. For Aim 3, the investigators will conduct non-inferiority analyses to compare pathogen density in ambient and cooled shipping conditions. The findings will provide valuable insights to clinics and laboratories regarding the reliability and acceptability of using home-collected sputum samples for microbiological evaluation. Ultimately, this project has the potential to introduce a non-invasive and minimally burdensome method for infection detection and diagnosis in people with CF.

ELIGIBILITY:
Inclusion Criteria:

* People with a diagnosis of cystic fibrosis (CF) based on CF Foundation (CFF) guidelines. The CFF guidelines consider a diagnosis of CF based on: (1) two known disease-causing CFTR mutations (based on historical genetic testing in clinical documentation or PortCF, the CFF patient registry), OR (2) sweat chloride 60 mmol/L (based on historical sweat chloride testing in clinical documentation or PortCF) and phenotypic findings consistent with cystic fibrosis in more than one organ system, OR (3) CFF accredited center physician diagnosis, based on clinical manifestations in the absence of two CFTR mutations with full gene mapping (based on historical genetic testing in clinical documentation or PortCF).
* Age 18 years old or greater
* People with the ability to comply with study visits and study procedures as judged by the investigator.

Exclusion Criteria:

* Solid organ transplant recipients, given the presence of immunosuppression.
* Those who are unable to tolerate sputum induction (hypertonic saline) or the inability to attempt sputum expectoration.
* Subjects who do not have access to a FedEx location or pick-up services will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with cystic fibrosis from three cystic fibrosis centers
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Pseudomonas aeruginosa positive culture | at baseline

SECONDARY OUTCOMES:
Culture-positive detection of Staphylococcus aureus, Burkholderia cepacia complex, Aspergillus fumigatus and other CF pathogens. | at baseline
Bacterial density in sputum measured by colony forming unit. | at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gina Hong, MD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - National Jewish Health, Denver, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No